CLINICAL TRIAL: NCT05326516
Title: AUGMENT-102: A Phase 1, Open-label, Dose-escalation Study to Evaluate Safety, Tolerability and Preliminary Anti-Leukemic Activity of SNDX-5613 in Combination With Chemotherapy in Patients With Relapsed/Refractory Leukemias Harboring Alterations in KMT2A/MLL, Nucleophosmin 1 (NPM1), and Nucleoporin 98 (NUP98) Genes
Brief Title: A Study of Revumenib in Combination With Chemotherapy in Participants With R/R Acute Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Syndax Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNDX-5613-0702
Expanded Access: NCT05918913 (No longer available)
Record Dates: First submitted 2022-03-23; First posted 2022-04-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Relapsed/Refractory Leukemias; Acute Lymphoblastic Leukemia; Acute Lymphocytic Leukemia; Mixed Phenotype Acute Leukemia; Acute Myeloid Leukemia; Acute Undifferentiated Leukemia
Keywords: SNDX-5613; AUGMENT; KMT2A/MLL Gene Rearrangement; Nucleophosmin 1 Mutation; NPM1; Nucleoporin 98; NUP98; Menin; Revumenib
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Biphenotypic, Acute; Leukemia, Myeloid, Acute | interventions — revumenib

STUDY DESIGN:
Intervention Model Description: The study will use a Bayesian optimal interval (BOIN) design to evaluate the doses and determine the maximum tolerated dose.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Revumenib and Chemotherapy Regimen 1 (Experimental): Participants with acute lymphoblastic leukemia/mixed phenotype acute leukemia (ALL/MPAL) will receive revumenib every 12 hours in combination with 2 treatment cycles of Chemotherapy Regimen 1.
  Interventions: Drug: Revumenib; Drug: Chemotherapy Regimen 1
- Revumenib and Chemotherapy Regimen 2 (Experimental): Participants with ALL/MPAL or acute myeloid leukemia (AML) will receive revumenib every 12 hours in combination with 2 treatment cycles of Chemotherapy Regimen 2.
  Interventions: Drug: Revumenib; Drug: Chemotherapy Regimen 2

INTERVENTIONS:
Drug: Revumenib — Participants will receive revumenib until meeting criteria for discontinuation.
  Other Names: SNDX-5613
Drug: Chemotherapy Regimen 1 — Participants will receive 2 treatment cycles of chemotherapy. During Cycle 1, participants will receive prednisone, vincristine, pegaspargase/calaspargase pegol-mknL, and daunorubicin. During Cycle 2, participants will receive etoposide and cyclophosphamide.
  Arms: Revumenib and Chemotherapy Regimen 1
Drug: Chemotherapy Regimen 2 — Participants will receive 2 treatment cycles of chemotherapy. During Cycles 1 and 2, participants will receive fludarabine and cytarabine.
  Arms: Revumenib and Chemotherapy Regimen 2

SUMMARY:
The purpose of this study is to determine the safety and tolerability of revumenib when given in combination with 2 different chemotherapy regimens in participants with relapsed/refractory acute leukemias harboring KMT2A rearrangement, KMT2A amplification, NPM1c, or NUP98r.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants must have documented relapsed or refractory (R/R) AML, ALL, or acute leukemias of ambiguous lineage (ALAL) including MPAL and acute undifferentiated leukemia (AUL) harboring KMT2A rearrangement, KMT2A amplification, NPM1c, or NUP98r.
* White blood count must be <25,000/microliter prior to the first dose of revumenib. Participants may receive cytoreduction per protocol prior to beginning revumenib.
* Eastern Cooperative Oncology Group performance status score 0-2 (if aged ≥18 years); Karnofsky Performance Scale of ≥50 (if aged ≥16 years and <18 years); Lansky Performance Score of ≥50 (if aged <16 years).
* Adequate liver, kidney, and cardiac function
* Participant must be taking 1 of the following medications for antifungal prophylaxis: itraconazole, ketoconazole, posaconazole, or voriconazole.
* A female of childbearing potential must agree to use a highly effective method of contraception or double barrier method from the time of enrollment through 120 days following the last study drug dose.

  * A male of childbearing potential must agree to use barrier contraception from the time of enrollment through 120 days following the last study drug dose.

Key Exclusion Criteria:

* Any unresolved ≥Grade 2 reversible toxicity from previous anticancer therapy except alopecia or Grade 2 neuropathy
* Graft-Versus-Host Disease (GVHD): Signs or symptoms of acute or chronic GVHD >Grade 0 within 4 weeks of enrollment. All transplant participants must have discontinued all systemic immunosuppressive therapy for at least 2 weeks and calcineurin inhibitors for at least 4 weeks prior to enrollment. Participants may be on physiological doses of steroids.
* Concurrent malignancy in the previous 2 years, with the exception of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (for example, breast carcinoma, cervical cancer in situ, melanoma in situ) treated with potentially curative therapy. Concurrent malignancy must be in complete remission or no evidence of disease during this timeframe. For participants with therapy-related leukemia, primary disease must be in remission for 1-year following completion of therapy.
* If the participant is known to be human immunodeficiency virus (HIV)-positive, the participant must have undetectable HIV viral load within the previous 6 months.
* Hepatitis B
* Hepatitis C
* Cardiac Disease:

  * Any of the following within the 6 months prior to study entry: myocardial infarction, uncontrolled/unstable angina, congestive heart failure (New York Heart Association Classification Class ≥II), life-threatening uncontrolled arrhythmia, cerebrovascular accident, or transient ischemic attack.
  * QTcF interval >450 milliseconds
* Any gastrointestinal (GI) issue of the upper GI tract that might affect oral drug absorption or ingestion (for example, gastric bypass, gastroparesis).
* Cirrhosis with a Child-Pugh score of B or C
* Down Syndrome
* Genetic syndromes: Bloom syndrome, ataxia-telangiectasia, Fanconi anemia, Kostmann syndrome, Shwachman syndrome, or any other known bone marrow failure syndrome.
* Participation in another therapeutic interventional clinical study within 28 days of starting revumenib.
* Radiation Therapy: within 60 days from prior total body irradiation, craniospinal radiation and/or ≥50% radiation of the pelvis, or within 14 days from local palliative radiation therapy (small port).
* Stem Cell Infusion or Donor Lymphocyte Infusion: within 60 days from hematopoietic stem cell transplantation and within 28 days from donor lymphocyte infusion without conditioning.
* Biologics (for example, monoclonal antibody therapy, bispecific antibodies, and antibody-drug conjugates): within 28 days or 5 half-lives, whichever is longer, since the completion of therapy with a biologic agent.
* Immunotherapy: within 42 days since tumor vaccines and checkpoint inhibitors, and within 21 days since receipt of chimeric antigen receptor therapy or other modified T-cell therapy.
* Hematopoietic Growth Factors: within 7 days since the completion of therapy with short-acting hematopoietic growth factors and within 14 days with long-acting growth factors.

Min Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-07-29 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Dose Limiting Toxicities From Revumenib | Day 1 through up to 30 days after last dose of study intervention
Number of Participants With Treatment-emergent Adverse Events | Day 1 through up to 30 days after last dose of study intervention

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of Revumenib | Predose through up to 6 hours postdose
Area Under The Plasma Concentration Versus Time Curve From Time 0 To t (AUC0-t) Of Revumenib | Predose through up to 6 hours postdose
Area Under The Concentration Versus Time Curve From Time 0 To 24 Hours (AUC0-24) Of Revumenib | Predose through up to 6 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Nicole McNeer, MD, PhD, Study Director — Syndax Pharmaceuticals
Locations (11):
- United States (10):
  - University of California, San Francisco (UCSF) Benioff Children's Hospital, San Francisco, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Children's Mercy Hospital, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - David H Koch Center for Cancer Care at Memorial Sloan Kettering Cancer Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Inc, Memphis, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Children's Cancer and Hematology Center, Houston, Texas
- Jewish General Hospital, Québec, Montreal, Canada

IPD SHARING:
Plan to Share IPD: No